CLINICAL TRIAL: NCT00805428
Title: Importance of CD4+CD25+ly in UC1. Investigation of Difference Between Blood Concentration IL 17, IL 33, Regulatory T ly in Patients With UC and Control Group
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Center, Split (Other)
Responsible Party: Jasna Ajdukovic, General practice
Other Study IDs: UC
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: control group
- patients with UC: patients with UC, without corticosteroid or immunosuppressive therapy

SUMMARY:
Mucosal inflammation in patients with UC is the result of immunosuppression disturbance because decreasing number of regulatory T ly and activation IL 17

ELIGIBILITY:
Inclusion Criteria:

* endoscopic confirmed diagnosis

Exclusion Criteria:

* corticosteroid or immunosuppressive therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with UC and control group
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2008-09

CONTACTS AND LOCATIONS:
Locations (1):
- Klinički bolnički centar Split, Split, Croatia